CLINICAL TRIAL: NCT02132637
Title: A Comparison of Pharmacodynamics When Receiving a Double Dose of Insulin Peglispro or Insulin Glargine in Patients With Type 2 Diabetes Mellitus: A Double-Blind, Crossover Design Study
Brief Title: A Study to Compare the Effect of a Double Dose of Two Long-acting Insulin Therapies in Participants With Type 2 Diabetes
Acronym: IMAGINE 8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14288; I2R-MC-BIDD (Other: Eli Lilly and Company); 2012-005174-56 (EudraCT Number)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — basal insulin peglispro; LY2605541; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Peglispro (Experimental): Standard dose of insulin peglispro administered subcutaneously (SQ) once daily for 4 weeks in one of two study periods. Double dose of insulin peglispro administered once, SQ on day 3 of the inpatient stay.
  Interventions: Drug: Insulin Peglispro
- Insulin Glargine (Experimental): Standard dose of insulin glargine administered subcutaneously (SQ) once daily for 4 weeks in one of two study periods. Double dose of insulin glargine administered once, SQ on day 3 of the inpatient stay.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Peglispro — Administered SQ
  Other Names: LY2605541
  Arms: Insulin Peglispro
Drug: Insulin Glargine — Administered SQ
  Arms: Insulin Glargine

SUMMARY:
The primary purpose of this study is to compare the effect of a double dose of a study drug known as insulin peglispro to a double dose of insulin glargine in participants who have type 2 diabetes. Participants will be treated with study insulin daily, in two 4-week study periods. Each participant will receive insulin peglispro during one treatment period and insulin glargine during the other treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM), based on the World Health Organization (WHO) classification, for ≥1 year.
* Use any type of basal insulin (except degludec), including once-or twice-daily human insulin neutral protamine Hagedom (NPH), insulin detemir, or insulin glargine.
* Have hemoglobin A1c (HbA1c) levels ≤9.0% according to local laboratory testing at screening.
* Have body mass index (BMI) ≤40.0 kilograms/square meter (kg/m^2).
* Have been treated with stable doses of insulin for at least 30 days before screening with:

  * Basal insulin with daily doses ±30% of mean during the last 4 weeks.
  * Doses of a basal insulin must be between 0.3 unit/kg/day and 1 unit/kg/day.
* If on metformin, thiazolidinediones (TZDs), sodium glucose co-transporter 2 (SGLT-2) inhibitors, or dipeptidyl peptidase (DPP4) inhibitors, must be on stable doses for the last 30 days.

Exclusion Criteria:

* Are using prandial, self-mixed, or premixed insulin. Participants using prandial insulin may be switched to everyday (qd) glargine if investigator judges that the participant will still meet fasting glucose requirements for randomization.
* Are using insulin pump therapy.
* Have excessive insulin resistance: Defined as >1.0 unit/kg/day as baseline treatment.
* If being treated with sulfonylureas (SUs) before screening, then must have SUs washed out between screening and randomization.
* Use any of these concomitant medications: morphine, codeine, antidiuretics, glucagon-like peptide-1 (GLP-1) receptor agonists (for example, exenatide, exenatide once weekly, lixisenatide or liraglutide), or pramlintide, used concurrently or within 90 days before screening.
* Have hypoglycemia unawareness, defined as confirmed by laboratory test results or by historical episodes of hypoglycemia <54 mg/dL (3.0 mmol/L) without symptoms.
* Have fasting hypertriglyceridemia >400 mg/dL (>4.5 mmol/L) at screening, as determined by the local laboratory.
* Have had any episode of severe hypoglycemia (defined by requiring assistance due to neurologically disabling hypoglycemia) within 6 months before entry into the study.
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control in the past 6 months.
* Have had a previous clinically significant episode of ketoacidosis as determined by the investigator (ketone bodies at fasting and without acidosis is acceptable) in the past 6 months.
* Have history of renal transplantation, are currently receiving renal dialysis, or have estimated Glomerular Filtration Rate (eGFR) <60 milliliters/minute.
* Have obvious clinical signs or symptoms of liver disease (excluding nonalcoholic fatty liver disease), acute or chronic hepatitis, nonalcoholic steatohepatitis, or elevated liver enzyme measurements.
* Have active or untreated malignancy, have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer) for less than 5 years, or are at increased risk for developing cancer or a recurrence of cancer in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Profil Institute for Clinical Research Inc, Chula Vista, California, United States
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Peglispro/Insulin Glargine: Standard dose of insulin peglispro administered subcutaneously (SQ) once daily for 4 weeks in the first study period. Double dose of insulin peglispro administered once, SQ on day 3 of the inpatient stay.
  Standard dose of insulin glargine administered subcutaneously (SQ) once daily for 4 weeks in the second study period. Double dose of insulin glargine administered once, SQ on day 3 of the inpatient stay.
- Insulin Glargine/Insulin Peglispro: Standard dose of insulin glargine administered subcutaneously (SQ) once daily for 4 weeks in the first study period. Double dose of insulin glargine administered once, SQ on day 3 of the inpatient stay.
  Standard dose of insulin peglispro administered subcutaneously (SQ) once daily for 4 weeks in the second study period. Double dose of insulin peglispro administered once, SQ on day 3 of the inpatient stay.
Period: Study Period 1
Arm/Group | Insulin Peglispro/Insulin Glargine | Insulin Glargine/Insulin Peglispro
Started | 34 | 34
Received at Least One Dose of Study Drug | 34 | 34
Completed | 33 | 30
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Physician Decision | 1 | 0
Period: Study Period 2 (Crossover)
Arm/Group | Insulin Peglispro/Insulin Glargine | Insulin Glargine/Insulin Peglispro
Started | 33 | 30
Completed | 31 | 29
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Peglispro/Insulin Glargine | Insulin Glargine/Insulin Peglispro | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.82 (8.06) | 57.74 (5.86) | 57.78 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 30 | 29 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 32 | 34 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10
  Germany | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Significant Hypoglycemia
Description: The percentage was calculated by dividing the number of participants with clinically significant hypoglycemia events defined as blood glucose <54 milligrams per deciliter (mg/dL) (3.0 millimole per liter [mmol/L]) or symptoms of severe hypoglycemia by the total number of participants analyzed, multiplied by 100.
Time Frame: Predose to 84 Hours Post Double Dose
Population: All randomized participants who received the double dose of study drug and had evaluable hypoglycemia data were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 61 | 62
percentage of participants | 6.6 | 35.5

2. Secondary Outcome: Percentage of Participants With Clinically Significant Hypoglycemia 12 Hours Post Double Dose
Description: The percentage was calculated by dividing the number of participants with clinically significant hypoglycemia events defined as blood glucose <54 mg/dL (3.0 mmol/L) or symptoms of severe hypoglycemia by the total number of participants analyzed, multiplied by 100.
Time Frame: Predose to 12 Hours Post Double Dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 61 | 62
percentage of participants | 1.6 | 22.6

3. Secondary Outcome: Percentage of Participants With Hypoglycemia
Description: The percentage was calculated by dividing the number of participants with hypoglycemia events defined as blood glucose ≤70 mg/dL (3.9 mmol/L) by the total number of participants analyzed, multiplied by 100.
Time Frame: Predose to 12 Hours Post Double Dose and 84 Hours Post Double Dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 61 | 62
percentage of participants
  12 Hours Post Double Dose | 19.7 | 64.5
  84 Hours Post Double Dose | 42.6 | 82.3

4. Secondary Outcome: Nadir Glucose
Description: Nadir glucose was defined as the lowest blood glucose for a participant with blood glucose ≤70 mg/dL (3.9 mmol/L). Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis including the following fixed effects: treatment, period, sequence, and baseline basal insulin dose stratification factor.
Time Frame: Predose to 84 Hours Post Double Dose
Population: All randomized participants who received the double dose of study drug and had blood glucose ≤70 mg/dL (3.9 mmol/L) during the first 84 hours after the double dose were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 26 | 51
mg/dL | 61.70 (1.36) | 55.93 (0.97)

5. Secondary Outcome: Time to the Nadir Glucose
Description: Nadir glucose was defined as the lowest blood glucose for a participant with blood glucose ≤70 mg/dL (3.9 mmol/L). The average time was calculated by dividing the sum of time from double dose to the nadir glucose for participants with blood glucose ≤70 mg/dL (3.9 mmol/L) by the number of participants with blood glucose ≤70 mg/dL (3.9 mmol/L) during the first 84 hours after the double dose.
Time Frame: Predose to 84 Hours Post Double Dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 26 | 51
hours | 35.92 (26.37) | 28.15 (23.46)

6. Secondary Outcome: Duration of Glucose ≤70 mg/dL
Description: The duration in minutes of each hypoglycemia episode with glucose ≤70 mg/dL (3.9 mmol/L) was calculated from start time to end time. The duration for a participant was the sum of the durations over the multiple hypoglycemia episodes. LS means were calculated using an MMRM analysis including the following fixed effects: treatment, period, sequence, and baseline basal insulin dose stratification factor.
Time Frame: Predose to 84 Hours Post Double Dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes per participant
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 61 | 62
Minutes per participant | 95.28 (37.57) | 362.26 (37.26)

7. Secondary Outcome: Fasting Blood Glucose
Description: Fasting blood glucose (FBG) was measured by self-monitored blood glucose. LS means were calculated by MMRM analysis with fixed effects of treatment, dosing day, sequence, period, interaction of treatment and dosing day, baseline basal insulin dose stratification factor, and baseline FBG.
Time Frame: Day 1, Day 2, and Day 3 Following Double Dose
Population: All randomized participants who received the double dose of study drug and had evaluable fasting blood glucose data were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 62 | 62
mg/dL
  Day 1: number analyzed (Participants) | 61 | 62
  Day 1 | 102.03 (2.90) | 85.61 (2.87)
  Day 2: number analyzed (Participants) | 62 | 61
  Day 2 | 100.94 (2.92) | 86.16 (2.91)
  Day 3: number analyzed (Participants) | 62 | 61
  Day 3 | 102.18 (2.99) | 86.27 (3.00)

8. Secondary Outcome: Pharmacodynamics: Three-Hour Postprandial Glucose Area Under the Concentration Time Curve (AUC)
Description: Glucose AUC within 3 hours after each meal assessed by the AUC of glucose from preprandial to 3 hours postprandial. LS means were calculated using an MMRM analysis including the following fixed effects: treatment, period, sequence, and baseline basal insulin dose stratification factor.
Time Frame: Preprandial to 3 Hours Postprandial during the day following the standard dose
Population: All randomized participants who received at least one dose of study drug and had evaluable glucose data were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL*h
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 62 | 63
mg/dL*h
  Breakfast | 633.50 (15.59) | 568.64 (15.51)
  Lunch | 566.00 (19.92) | 568.20 (19.84)
  Dinner: number analyzed (Participants) | 62 | 62
  Dinner | 564.68 (15.95) | 577.46 (15.95)

9. Secondary Outcome: Pharmacodynamics: Three-Hour Postprandial Glucose Area Under the Concentration Time Curve (AUC) Excursion
Description: Glucose AUC excursion within 3 hours after each meal assessed by the AUC of adjusted glucose (= observed glucose - preprandial glucose) from preprandial to 3 hours postprandial. LS means were calculated using an MMRM analysis including the following fixed effects: treatment, period, sequence, and baseline basal insulin dose stratification factor.
Time Frame: Preprandial to 3 Hours Postprandial during the day following the standard dose
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mg/dL*h
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 62 | 63
mg/dL*h
  Breakfast | 266.33 (12.04) | 270.32 (11.98)
  Lunch | -2.38 (11.42) | 36.92 (11.34)
  Dinner: number analyzed (Participants) | 62 | 62
  Dinner | 134.40 (10.20) | 150.23 (10.20)

10. Secondary Outcome: Beta Cell Function
Description: Beta cell function assessed by the change between pre meal tolerance test and 30 minutes post meal tolerance test in C-peptide corrected insulin/Glucose (ΔC-peptide corrected insulin/ΔGlucose). LS means were calculated using an MMRM analysis including the following fixed effects: treatment, period, sequence, and baseline basal insulin dose stratification factor.
Time Frame: 0-30 minutes during the meal tolerance test on the day following the standard dose
Population: All randomized participants who received at least one dose of study drug and had evaluable ΔC-peptide data were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 64 | 67
mmol/L | 88.65 (8.43) | 103.62 (8.32)

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug.
Arm/Group | Insulin Peglispro | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 2/64 | 1/67
Other Adverse Events (participants affected / at risk) | 31/64 | 26/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=64) | Insulin Glargine (N=67)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=64) | Insulin Glargine (N=67)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (6)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 11 (16) | 7 (7)
Irritability (General disorders) | 1 (1) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days